CLINICAL TRIAL: NCT05336110
Title: Assessment of the Impact of the Postponement of Surgery on the Postoperative Morbidity After Sars-cov-2 Infection in 2022
Brief Title: Impact of the Postponement of Surgery on Postoperative Morbidity After Sars-cov-2 Infection
Acronym: DROMIS-22
Status: Completed | Type: Observational
Sponsor: Société Française d'Anesthésie et de Réanimation (Other)
Responsible Party: Sponsor
Other Study IDs: DROMIS-22 / 2022-01; 2022-A00228-35 (Other: ID-RCB)
Record Dates: First submitted 2022-03-21; First posted 2022-04-20 (Actual); Last update posted 2022-07-18 (Actual); Status verified 2022-07

CONDITIONS: SARS CoV 2 Infection
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient with a positive preoperative SARS-CoV-2 test: Patient with a positive preoperative SARS-CoV-2 test
  Interventions: Other: Postponing surgery

INTERVENTIONS:
Other: Postponing surgery — Postponing surgery for patients with Sars-cov-2 infection

SUMMARY:
The deployment of vaccination against SARS-CoV-2 from 2021 led to a modification in June 2021of previous recommendations concerning the postponing scheduled surgery suggesting local adaptations of this delay if epidemic developments appear. Today, the evolutions of the pandemic make these recommendations obsolete and impose the updating of the data produced during the first epidemic wave of 2020. Among these evolutions, the two most important are the existence of a large vaccination coverage on the one hand and the emergence of variants of lesser severity on the other hand

DETAILED DESCRIPTION:
Previous studies performed during the first COVID-19 epidemic wave in the first half of 2020 led to the recommendation, after taking into account the individual risk-benefit balance, of postponing scheduled surgery for ideally at least 6 completed weeks in a patient with a positive preoperative SARS-CoV-2 PCR.

The deployment of vaccination against SARS-CoV-2 from 2021 led to a modification of these recommendations in June 2021 suggesting local adaptations of this delay if epidemic developments appear. Today, the evolutions of the pandemic make these recommendations obsolete and impose the updating of the data produced during the first epidemic wave of 2020. Among these evolutions, the two most important are the existence of a large vaccination coverage on the one hand and the emergence of variants of lesser severity on the other hand

ELIGIBILITY:
Inclusion Criteria:

* Adult patients,
* Surgery performed in the operating room under general or locoregional anesthesia.
* Result of the preoperative SARS-COV-2 diagnostic test available on the day of the procedure or within 48 hours of the surgery.
* Emergency or scheduled surgery
* All surgical indications will be eligible with the exception of certain surgeries

Exclusion Criteria:

* Minor patient
* Pregnant patient
* Surgery or an intervention performed outside the operating room
* Patient operated under sedation alone,
* Patient under guardianship or curatorship
* Patient without social protection
* Patient previously included in this study
* Patient without preoperative COVID-19 status on day of surgery and not diagnosable within 48 postoperative hours
* Patient whose immediate postoperative follow-up is planned in a structure other than those where the inclusion was made

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient going to have surgery
Sampling Method: Probability Sample
Enrollment: 5189 (Actual)
Dates: Start 2022-03-14 (Actual); Primary Completion 2022-05-13 (Actual); Study Completion 2022-05-13 (Actual)

PRIMARY OUTCOMES:
Composite endpoint, that consist of respiratory morbidity associated with occurrence of respiratory events and use or prolongation of mechanical ventilation. | up to 30 postoperative days.
  The primary endpoint will be a composite endpoint, that consist of respiratory morbidity associated with occurrence of pneumonia (bacterial or viral), acute respiratory distress, symptomatic pulmonary embolism (i.e. having led to a diagnostic procedure and a treatment), and postoperative prolongation of mechanical ventilation or the use of unscheduled, during the postoperative hospital stay and within the limit of 30 postoperative days.

SECONDARY OUTCOMES:
Secondary Outcome Measures include hospital mortality, | up to 30 postoperative days.
  The secondary endpoints will be the hospital mortality (number of death during hospitalization)
Secondary Outcome Measures include mortality at D30, | up to 30 postoperative days.
  The secondary endpoints will be the mortality at D30 (number of death since surgery until Day 30);
Secondary Outcome Measures include the occurrence of a deep vein thrombosis, | up to 30 postoperative days.
  The secondary endpoints will be the number of occurrence of a deep vein thrombosis (excluding pulmonary embolism),
Secondary Outcome Measures include non-respiratory infection and septic shock, | up to 30 postoperative days.
  The secondary endpoints will be the numberof non-respiratory infection or septic shock during the post-operative hospital stay and within the limit of postoperative 30 days.
Secondary Outcome Measures include non-respiratory infection or septic shock, | up to 30 postoperative days.
  The secondary endpoints will be the number of non-respiratory infection or septic shock during the post-operative hospital stay and within the limit of postoperative 30 days.
Secondary Outcome Measures include length of hospital stay and length of critical care stay. | up to 30 postoperative days.
  The secondary endpoints will be the length of hospital stay, length of critical care stay (if hospitalization in critical care).
Secondary Outcome Measures include the need for re-hospitalization during the first 30 days after surgery | up to 30 postoperative days.
  The secondary endpoints will be the need for re-hospitalization during the first 30 days after surgery (number of patients with re-hospitalization)

CONTACTS AND LOCATIONS:
Overall Officials: Marc GARNIER, MD, Principal Investigator — HOPITAL TENON - PARIS
Locations (40):
- France (40):
  - CHU d'Amiens, Amiens
  - CHU d'Angers, Angers
  - CH Victor Dupouy, Argenteuil
  - Cinique Belharra, Bayonne
  - CH de Blois, Blois
  - CHU de Brest - la Cavale Blanche, Brest
  - HIA Clermont Tonnerre, Brest
  - CHU de Caen - Anesthésie Réanimation, Caen
  - CHU de Caen, Caen
  - CH Charleville Mézière - CH Intercommunal Nord Ardennes, Charleville-Mézières
  - AP-HP - Hôpital Beaujon, Clamart
  - Hôpital Antoine Béclère, Clamart, Clamart
  - CHU Clermont-Ferrand, Clermont-Ferrand
  - Centre Hospitalier Sud Francilien, Corbeil-Essonnes
  - CHU Grenoble-Alpes, La Tronche
  - CHU de Lille - hôpital Claude Huriez, Lille
  - Hôpital E. Herriot - Hospices Civils de Lyon, Lyon
  - CHU La Timone - Marseille, Marseille
  - Hôpital Nord, Marseille, Marseille
  - Clinique du Sport de Bordeaux Mérignac, Mérignac
  - CHU de Nantes, Nantes
  - Hopital Tenon, Paris
  - AP-H P - Hôpital Lariboisière, Paris
  - AP-HP - Groupe Hospitalier Pitié-Salpêtrière (bloc central), Paris
  - AP-HP - Groupe Hospitalier Pitié-Salpêtrière, Paris
  - AP-HP - Hôpital Bichat, Paris
  - AP-HP - Hôpital Saint-Antoine, Paris
  - AP-HP - Hôpital Saint-Louis, Paris
  - Clinique Drouot Rémusa, Paris
  - Clinique Saint Jean de Dieu, Paris
  - Centre Henri Becquerel, Rouen
  - CHU Sud Réunion (Saint-Pierre), Saint-Pierre
  - CHU Strasbourg- Hautepierre, Strasbourg
  - CHU de Toulouse -Hôpital Purpan, Toulouse
  - CHU de Toulouse -Hôpital rangueil, Toulouse
  - Clinique Pasteur, Toulouse, Toulouse
  - CHRU de Tours - Hôpital Trousseau, Tours
  - Institut de Cancérologie de Lorraine, Vandœuvre-lès-Nancy
  - Centre Gustave Roussy, Villejuif
  - Polyclinique de Villeneuve Saint Georges, Villeneuve-Saint-Georges